CLINICAL TRIAL: NCT00165035
Title: Multi-Center, Single-Blind, Two-Arm, Randomized, Controlled, Non Inferiority Trial of the Conor CoStar Paclitaxel-Eluting Coronary Stent System vs the TAXUS DES in Patients With De Novo Lesions of the Native Coronary Arteries
Brief Title: Cobalt Chromium Stent With Antiproliferative for Restenosis II Trial (COSTAR II)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cordis US Corp. (Industry)
Collaborators: Conor Medsystems (Industry)
Responsible Party: Mitch W Krucoff, MD, Principal Investigator, Duke University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: COSTAR II
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2011-08-04 (Estimated); Status verified 2011-08

CONDITIONS: Coronary Disease
Keywords: Percutaneous coronary intervention (PCI); Drug eluting stent (DES)
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): CoStar™ Paclitaxel-Eluting Coronary Stent, a reservoir based DES
  Interventions: Device: CoStar Paclitaxel Drug Eluting Coronary Stent System
- 2 (Active Comparator): TAXUS™ Express2™ Paclitaxel-Eluting Coronary Stent
  Interventions: Device: TAXUS™ Express2™ Paclitaxel-Eluting Coronary Stent

INTERVENTIONS:
Device: CoStar Paclitaxel Drug Eluting Coronary Stent System — Drug eluting stent
  Arms: 1
Device: TAXUS™ Express2™ Paclitaxel-Eluting Coronary Stent — Drug eluting stent
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of the investigational stent CoStar™ Paclitaxel-Eluting Coronary Stent- a reservoir based DES system in comparison to a surface coated DES stent (TAXUS™ Express2™ Paclitaxel-Eluting Coronary Stent) in the treatment of single-vessel (one blood vessel) and multi-vessel (two or three blood vessels) coronary artery disease.

DETAILED DESCRIPTION:
Non -inferiority in 8-month Major Adverse Cardiac Events (MACE) and in-segment late lumen loss at 9 months between the CoStar™ Paclitaxel-Eluting Coronary Stent System and the TAXUS™ Express2™ Drug Eluting Coronary Stent System for the treatment of a single de novo lesion per vessel in patients with single and multi-vessel coronary disease.

ELIGIBILITY:
Inclusion Criteria:

General Inclusion Criteria:

* Eligible for percutaneous coronary intervention (PCI)
* Documented stable or unstable angina pectoris (Class I, II, III or IV), documented ischemia, or documented silent ischemia
* Documented LVEF ≥25% within the last 6 weeks.
* Eligible for coronary artery bypass graft surgery (CABG)

Exclusion Criteria:

General Exclusion Criteria:

* Known sensitivity to paclitaxel or polymeric matrices: Translute or PLGA.
* Planned treatment with any other PCI device in the target vessel(s).
* MI within 72 hours prior to the index procedure
* Patient is in cardiogenic shock
* Cerebrovascular Accident (CVA) within the past 6 months
* Acute or chronic renal dysfunction (creatinine >2.0 mg/dl or >150 µmol/L)
* Contraindication to ASA or to clopidogrel
* Thrombocytopenia
* Active GI bleeding within past three months
* Known allergy to stainless steel or cobalt chromium
* Any prior true anaphylactic reaction to contrast agents
* Patient is currently taking colchicine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1701 (Actual)
Dates: Start 2005-05; Primary Completion 2007-01 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
MACE defined as a composite of target vessel revascularization, new myocardial infarction (MI), or cardiac death | 8 months
In-segment late lumen loss | 9 months

SECONDARY OUTCOMES:
Device, lesion and procedure success | At procedure or hospital discharge
Incidence of MACE | 30 days, 9 months and 12 months
Coronary angiography in the angiographic cohort | 9 months
Target lesion revascularization | 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Dean J Kereiakes, MD, Principal Investigator — The Christ Hospital, Cincinnati, Ohio; Mitchell W Krucoff, MD, Principal Investigator — Duke University Medical Center, Durham, NC
Locations (2):
- United States (2):
  - Duke University Medical Center, Durham, North Carolina
  - Christ Linder, Cincinnati, Ohio

REFERENCES:
- [Result] Kereiakes DJ, Petersen JL, Batchelor WB, Fitzgerald PJ, Mehran R, Lansky A, Tsujino I, Schofer J, Dubois C, Verheye S, Cristea E, Garg J, Wijns W, Krucoff MW. Clinical and angiographic outcomes in diabetic patients following single or multivessel stenting in the COSTAR II randomized trial. J Invasive Cardiol. 2008 Jul;20(7):335-41. PMID 18599890
- [Result] Krucoff MW, Kereiakes DJ, Petersen JL, Mehran R, Hasselblad V, Lansky AJ, Fitzgerald PJ, Garg J, Turco MA, Simonton CA 3rd, Verheye S, Dubois CL, Gammon R, Batchelor WB, O'Shaughnessy CD, Hermiller JB Jr, Schofer J, Buchbinder M, Wijns W; COSTAR II Investigators Group. A novel bioresorbable polymer paclitaxel-eluting stent for the treatment of single and multivessel coronary disease: primary results of the COSTAR (Cobalt Chromium Stent With Antiproliferative for Restenosis) II study. J Am Coll Cardiol. 2008 Apr 22;51(16):1543-52. doi: 10.1016/j.jacc.2008.01.020. PMID 18420096